CLINICAL TRIAL: NCT01327144
Title: A Prospective, Randomized, Multicenter Study of the Efficacy and Safety of Famciclovir 500 mg Comparing To Aciclovir 400mg in Patients With Herpes Zoster
Brief Title: Efficacy of Oral Famciclovir Versus Aciclovir Treatment in Patients With Herpes Zoster
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: F500EMS1010
Record Dates: First submitted 2011-03-30; First posted 2011-04-01 (Estimated); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster | interventions — Famciclovir; Acyclovir

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Famciclovir 500mg (Experimental): 1 tablet each 8 hours for 7 days
  Interventions: Drug: Famciclovir
- Aciclovir 400mg (Active Comparator): 2 tablets of Aciclovir 400 mg each 4 hours for 7 days
  Interventions: Drug: Aciclovir

INTERVENTIONS:
Drug: Famciclovir — Famciclovir 500 mg- 1 tablet each 12 hours for 7 days
  Arms: Famciclovir 500mg
Drug: Aciclovir — Aciclovir 400 mg- 02 tablets each 4 hours for 7 days
  Arms: Aciclovir 400mg

SUMMARY:
Herpes Zoster is an infection that affects part of the nervous system caused by Varicella Zoster Virus. Herpes Zoster manifests as vesicular eruption in the dermatome, often associated with significant pain.

There are effective oral prescription antiviral medicines available to reduce the discomfort of symptoms as famciclovir and aciclovir.

This is a phase III, multicenter, randomized, parallel-group study to compare the efficacy and safety of treatment with Famciclovir (500 mg) comparing to Aciclovir (400 mg) in patients with Herpes Zoster.

DETAILED DESCRIPTION:
Study Design

* single blind study, prospective, parallel group, intent to treat trial
* Experiment duration: 7 days
* 2 visits (days 0, and 7)
* Reduction of symptoms
* Adverse events evaluation

ELIGIBILITY:
Inclusion Criteria:

* Patients must be able to understand the study procedures, agree to participate and give written consent.
* Patients with clinical diagnosis of Herpes Zoster;
* Score higher than 4 for at least for 2 symptoms of Herpes Zoster;
* Negative pregnant urine test

Exclusion Criteria:

* Pregnancy or risk of pregnancy.
* Lactation
* Any pathology or past medical condition that can interfere with this protocol.
* Non-steroidal anti-inflammatory drug , hormonal anti-inflammatory or immunosuppressive drugs (in the last 30 days and during the study);
* Patients with immunodeficiency and/or immunosuppressive disease;
* Hypersensitivity to components of the formula;
* Other conditions deemed reasonable by the medical investigator as to the disqualification of the individual from study participation.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 177 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2017-05 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
For efficacy evaluation, a visual analogue scale (VAS) will be used to detect the improvement of symptoms | day 7
  Symptoms evaluated: pain, injury, loss of sensation, burning and itching

SECONDARY OUTCOMES:
Safety will be evaluated by the adverse events occurrences | day 7
  Adverse events will be collected and followed in order to evaluate safety and tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Joyce Silva, MD, Study Director — EMS
Locations (5):
- Brazil (5):
  - Centro de Medicina Reprodutiva Dr Carlos Isaia Filho, Porto Alegre, Rio Grande do Sul
  - Loema, Campinas, São Paulo
  - Allergisa, Campinas, São Paulo
  - CECIP Centro de Estudos Clínicos do Interior Paulista, Jaú, São Paulo
  - Afip - Associacao Fundo de Incentivo A Pesquisa, São Paulo, São Paulo

REFERENCES:
- [Result] Pott Junior H, de Oliveira MFB, Gambero S, Amazonas RB. Randomized clinical trial of famciclovir or acyclovir for the treatment of herpes zoster in adults. Int J Infect Dis. 2018 Jul;72:11-15. doi: 10.1016/j.ijid.2018.04.4324. Epub 2018 May 7. PMID 29746903